CLINICAL TRIAL: NCT05943275
Title: Validation of a Magnetic Sensor for the Non-invasive Measurement of Jugular Venous and Radial Arterial Pressure in Patients During Cardiac Catheterization
Brief Title: Magnetic Sensor Validation of Hemodynamic Non-invasive Measurements Pressure During Cardiac Catheterization
Acronym: CapMag
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL21_0595; 2022-A00775-38 (Other: IDRCB)
Record Dates: First submitted 2023-06-23; First posted 2023-07-13 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-07

CONDITIONS: Complex Congenital Heart Disease; Chronic Right Heart Failure
Keywords: Non-invasive venous pressure measurement

STUDY DESIGN:
Intervention Model Description: comparison between two measurement methods, one of which serves as a reference in a single group of patients patients, without randomization, prospective and monocentric. This is a proof-of-concept pilot study. concept.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with an indication for right heart catheterization (Other): During the preparation of the subject on the cardiac catheterization table, a person specifically trained to the measurements of the medical device under test will be dedicated to this study. Once the skin has been cleaned with alcohol the device (magnet and micro-sensor encapsulated in the plastic support) will be placed on the subject's uninjured skin of the subject, on the path of the jugular vein. A second device will be placed at the level of the radial artery radial artery with the help of a bracelet. The signals will be recorded and observed on a screen for the duration of the invasive hemodynamic measurements, i.e. approximately 15 minutes.
  Interventions: Device: Magnetic sensor

INTERVENTIONS:
Device: Magnetic sensor — During the right heart catheterization procedure, measurement of hemodynamic pressures by the non-invasive experimental method (Magnetic sensor) and the invasive control method

SUMMARY:
Follow-up of patients with complex congenital heart disease (CHD) usually involves ultrasound imaging or even MRI or CT scans of the heart and stress testing. But these examinations can be challenged in terms of their sensitivity. Thus, the development of non-invasive jugular venous and radial arterial pressure sensors, reflecting the hemodynamic function of the right heart, would be very useful to the clinician responsible for early detection of a deficit in right ventricular function.

DETAILED DESCRIPTION:
Among the 1% of live births with congenital heart disease, 20% have complex congenital heart disease (CHD). Their life expectancy, initially low, is constantly improving due to diagnostic, follow-up and therapeutic advances, particularly surgical. The pediatric population surviving the neonatal period is increasingly high and the number of people reaching adulthood has even exceeded the pediatric population for the last 3 years, a number that puts adult cardiologists in difficulty as they have little knowledge of the natural history of these pathologies. Indeed, it is difficult to predict or diagnose early decompensation or deterioration of cardiac function, especially for those affecting right heart function, because the anatomic and hemodynamic particularities of these CHDs make the usual functional exploration parameters not very sensitive. Indeed, the dysfunction of ventricular function is progressive and these patients remain asymptomatic for a long time and then decompensate suddenly. The late symptoms and the anatomic difficulty in adapting paraclinical criteria used for morphologically normal hearts explain their difficult interpretation and a delay in management. The current evaluation of these CHDscombining ultrasound imaging or even MRI or cardiac CT and stress testing is often flawed in terms of their sensitivity, because of the anatomic geometric complexity of these heart diseases.

Thus, the development of a non-invasive jugular venous pressure sensor, reflecting the hemodynamic function of the right heart, would be very useful to the clinician responsible for the follow-up of subjects with CHD, in order to detect early a deficit in right ventricular function.

F. Terki and H. Tran of the DynaCar team "Dynamics of cardiac couplings" of the Laboratory of Physiology Experimental Medicine (PhyMedExp), have developed an innovative medical detection device in partnership with the Laboratory of Coordination Chemistry LCC of the CNRS of Toulouse (A. Bousseksou) and the company eV-technologies (S. Wane and H. Tran), allowing to measure this jugular venous pressure by simple apposition of this one on the vein. A small magnet of 1cm X 1cm is placed beside the sensor. The very weak magnetic field of this magnet (0,02 Tesla) will generate a voltage at the terminals of the micro-sensor placed just beside. This voltage will reflect the pressure force related to the blood flow circulating in the cardiovascular network and give information on the heartbeat by magnetic measurements. The magnet and the micro-sensor are encapsulated in a plastic support of 3cm X1 cm and clipped on a flexible bracelet that can be affixed to the neck.

The magnetic field of the magnet used is of the order of magnitude of that of the fridge magnets (0.02 Tesla). It is therefore not harmful. It is 75 times weaker than that used in MRI (1.5T).

This device does not require the use of contrast agents, no patch and no adhesive product and is without direct contact with the skin.

The signals detected by the microchip (microsensor) are then transmitted to a tablet or laptop computer via a wired USB connection. A second sensor will be positioned on the radial artery through a bracelet placed around the wrist. Thus a magnetic arterial measurement will be simultaneously recorded.

It is therefore proposed that this magnetic sensor, affixed to the jugular vein, which empties into the right atrium, has the same sensitivity as the bloody measurement of central venous pressure. For that purpose, in a first study, the research team want to compare, during a right catheterization, the blood venous pressure curve, which is the reference method, with the one obtained by the innovative magnetic sensor. Indeed, before evaluating the interest of this medical device on patients with a dysfunction of the cardiac pump, the sensitivity of the measurements obtained in subjects who will benefit from an invasive hemodynamic evaluation during their follow-up must be validated, which will allow us to obtain a reference measurement.

The technology proposed in this study is totally innovative. It is based on the measurement of the magnetic field generated by the blood fluid during its passage in a vessel, which is detected by a micro-sensor placed on the skin. Although the structure and measurement principle are completely innovative for this study, magnetic ultrasensitivity has been demonstrated. Validation of the sensitivity of these sensors to non-invasively detect variations in venous pressure at the jugular vein will allow the future development of non-invasive miniature 'smart devices' with very low energy consumption (80 microWatt) and high early prognostic value in relation to right heart failure, allowing the refinement of monitoring and re-evaluation of therapeutic management of patients with CHD. These devices will be developed, characterized, tested and deployed in Occitania. The synergy between academic (University of Montpellier, CNRS Toulouse, INSERM, CHUM) and industrial (eV-Technologies) actors will ensure that the entire value chain from the development of the microsensors to the acceleration of their valorization and technology transfer will be anchored in Occitanie.

ELIGIBILITY:
Inclusion Criteria:

* Patient who receives a right-sided catheterization
* Age ≥ 18 years
* Informed consent

Exclusion Criteria:

* Patient with a metal implant near the area of use of the device
* Pregnant or breastfeeding woman
* Patient unwilling or unable to sign consent: patient under guardianship or conservatorship, mentally retarded, dementia, language barrier
* Patient not affiliated to a social security system
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Estimate the concordance between the mean peak atrial pressure values measured by the two methods (invasive and magnetic sensor) over a 15-minute period. | Baseline
  Average value of the atrial peak pressure measured by both methods (invasive and magnetic sensor) over a 15-minute period.

SECONDARY OUTCOMES:
Assess whether there is an overlap between the jugular venous pressure curve obtained with a magnetic sensor and the invasive central venous pressure curve | baseline
  Concordance test between the average of the parameters describing the two pressure curves measured with the two methods (invasive and magnetic sensor) over a period of 15 minutes.
  Value of the peak pressure for the ventricular contraction (c wave)
Assess whether there is an overlap between the jugular venous pressure curve obtained with a magnetic sensor and the invasive central venous pressure curve (atrial filling) | baseline
  Concordance test between the average of the parameters describing the two pressure curves measured with the two methods (invasive and magnetic sensor) over a period of 15 minutes.
  Value of the peak pressure for the atrial filling (v wave)
Assess whether there is an overlap between the jugular venous pressure curve obtained with a magnetic sensor and the invasive central venous pressure curve (Area under the pressure curve during a cardiac revolution) | baseline
  Concordance test between the average of the parameters describing the two pressure curves measured with the two methods (invasive and magnetic sensor) over a period of 15 minutes.
  Value of the peak pressure for the Area under the pressure curve during a cardiac revolution.
Evaluate whether there is an overlap, during a simultaneous measurement, between the jugular venous pressure curve and the radial arterial pressure curve obtained with a magnetic and the radial arterial pressure curve obtained with a magnetic sensor | baseline
  visual identification of two pressure peaks with the presence of a cataclysmic incisure between systole and diastole on the blood pressure curve measured at the radial artery with the magnetic sensor.
To evaluate the safety of measuring jugular venous pressure or radial arterial pressure with a magnetic sensor in patients. | Baseline
  Collection of undesirable effects experienced by the patient during the installation of magnetic sensors during the measurement of venous pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Quentin DELBAERE, MD, Study Director — CHU de Montpellier
Locations (1):
- CHU de Montpellier Département de Cardiologie Hôpital Arnaud de Villeneuve, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided